CLINICAL TRIAL: NCT00032695
Title: Treatment of AIDS Vacuolar Myelopathy With Methionine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS035745 (NIH)
Record Dates: First submitted 2002-03-28; First posted 2002-03-29 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2005-11

CONDITIONS: Myelopathy; AIDS-Myelopathy; AIDS Vacuolar Myelopathy
Keywords: myelopathy; AIDS-myelopathy; AIDS vacuolar myelopathy; methionine
MeSH Terms: conditions — Spinal Cord Diseases | interventions — Methionine

INTERVENTIONS:
Drug: methionine

SUMMARY:
The purpose of this study is to determine whether methionine, an amino acid present in low doses in the normal diet, can improve myelopathy or stop its progression.

DETAILED DESCRIPTION:
Myelopathy is usually a late complication of AIDS, and until recently its symptoms were rarely recognized, masked by the general state of disability or the presence of other neurological complications. With prolonged survival and improved quality of life of HIV-infected patients, myelopathy is increasingly becoming a common source of disability. The cause of AIDS-myelopathy is unknown, but it is probably an indirect effect of the long-term presence of the HIV virus in the nervous system rather than the result of a direct infection. The purpose of this study is to determine whether methionine, an amino acid present in low doses in the normal diet, can improve myelopathy or stop its progression.

ELIGIBILITY:
Between 18 and 80 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Rocco, MD, Principal Investigator
Locations (1):
- Beth Israel Medical Center, New York, New York, United States